CLINICAL TRIAL: NCT06868966
Title: Implications of Myelin in Executive Control in Adolescence and Early Adulthood
Acronym: MYELEX
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D23-P028
Record Dates: First submitted 2024-07-11; First posted 2025-03-11 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Myelex study is a fundamental research study that aims to better understand how the brain functions and develops. The objective of this study is to better understand the role of myelin, a sheath that surrounds nerve fibers and determines the speed of information propagation in the brain, in cognitive functioning during development in adolescents and young adults. investigator use Magnetic Resonance Imaging (MRI) because this method allows us to study the anatomy and functioning of the brain in a non-invasive (no injection) and painless manner. investigator focus on cognitive control, a set of cognitive functions in the prefrontal cortex, at the front of the brain, that enable the use of the best strategies on a case-by-case basis to solve problems effectively. These functions are closely associated with academic and professional success and develop late, continuing until early adulthood. The goal of this project is simple: to measure the myelin of nerve fibers using MRI and to evaluate the link with the development of cognitive control. Each participant will undergo an MRI examination and cognitive assessments. The study takes place at the Clinical Research Center of GHU Paris and lasts a total of 3.5 hours, including reception, setup, MRI recording, and the completion of a series of cognitive tasks.

DETAILED DESCRIPTION:
Selection visit

* Call for participants for pre-selection
* Sending of information forms by mail
* Making an appointment for the inclusion visit Inclusion visit at GHU Paris.
* Information on the modalities, constraints and foreseeable risks of the study
* Collection of informed consent
* Verification of inclusion/non-inclusion criteria
* Clinical examination: o Verification of medical history and drug treatments

  * Psychiatric pathology in first-degree relatives
  * Consumption of toxic substances (nicotine, alcohol, cannabis, etc.)
  * Manual lateralization will be assessed by the score on the Edinburgh questionnaire (Oldfield, 1971)
  * Blood sample to measure pubertal hormones (testosterone, estradiol and progesterone levels)
* Collection of main medical history and concomitant treatments
* Explanation of study procedures
* MRI examination
* Cognitive assessment

ELIGIBILITY:
Inclusion Criteria:

* Male or female; Subject aged 10 to 25 years; Right-handed preference; Subject, or legal representative, who has given consent to participate; Native language: French; Subject affiliated with a social security system; Having signed their consent to participate (and their legal representative if applicable), subjects and parents have read the information letter and given their free and informed consent. In cases where only one parent gives consent (for minors), this must be justified (such as no contact with the other parent for over a year).

Exclusion Criteria:

* Not corresponding to the targeted age range;
* Subject with contraindications to an MRI examination (pacemaker or neurosensory stimulator or implantable defibrillator, cochlear implants, ferromagnetic foreign bodies in the eyes or brain near neural structures, metal prostheses, patient agitation: non-cooperative or agitated patients, minors, claustrophobic subjects, pregnant women, ventriculoperitoneal neurosurgical shunt valves, dental braces);
* Subject with chronic alcohol or drug use;
* Abuse or dependence on substances (except nicotine) or toxic substances for more than 5 years or having led to comas (overdoses);
* Subject with sudden-onset cognitive disorders that could indicate a stroke; a history of head trauma with loss of consciousness for more than 1 hour, or encephalitis;
* Subject with chronic neurological, psychiatric, endocrine, hepatic, or infectious conditions;
* Subject with a history of major illness (diabetes, chronic lung disease, severe cardiac, metabolic, hematological, endocrine, or immunological disorder, cancer);
* Subject on medication: taking medications likely to interfere with brain imaging measurements (psychotropics, anxiolytic hypnotics, neuroleptics, anti-Parkinsonians, benzodiazepines, steroidal anti-inflammatories, antiepileptics, central analgesics, and muscle relaxants);
* Color blindness;
* Inability to comply with the study for geographical or psychiatric reasons;
* Tattoo incompatible with MRI;
* Cerebral palsy;
* Fine motor skills disorder;
* Pregnant women at the time of inclusion;
* Adult subjects under legal protection or unable to give consent (article L.1121-8 of the French Public Health Code) (under guardianship or curatorship);
* Children and parents under legal protection measures

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy adolescent and adult volunteers aged 10 to 25 years with no contraindications for an MRI examination.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Myelin | Day 1
  Myelin Levels : Regional variations of Fractional Anisotropy (FA)

SECONDARY OUTCOMES:
Working Memory | Day 1
  Spatial Span from CANTAB
  - Units on a Scale
Inhibitory skills | Day 1
  Stop Signal Task from CANTAB and CHEXI, TEXI and ADEXI self-questionnaires
  - Units on a Scale
Planning skills | Day 1
  One Touch Stockings of Cambridge - Units on a Scale
Decision-making and risk-taking | Day 1
  Cambridge Gambling Task from CANTAB - Units on a Scale
Reading skills | Day 1
  Text, word and pseudoword reading and metaphonology from EVALEO 6-15/ECLA16+/EXALANG - Units on a Scale
IQ | Day 1
  Raven's Standard Progressive Matrices (SPM) - Units on a Scale
Reasoning | Day 1
  Cognitive Reasoning Task - Units on a Scale
Social Cognition | Day 1
  Tom-15 task - Units on a Scale
Visuospatial attention | Day 1
  Multiple Object Tracking task from CRAB - Units on a Scale
Wellbeing questionnaire | Day 1
  KIDSCREEN 27 for minor participants and SF-36 for adults - Units on a Scale
Behavior questionnaire | Day 1
  BIS/BAS scales - Units on a Scale
Self-regulation questionnaire | Day 1
  DERS-F - Units on a Scale
Demographics questionnaire | Day 1
  Age, sex, level of studies, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Ste Anne, Paris, France